CLINICAL TRIAL: NCT02143830
Title: A Phase II Trial of HSCT for the Treatment of Patients With Fanconi Anemia Lacking a Genotypically Identical Donor, Using a Risk-Adjusted Chemotherapy Only Cytoreduction With Busulfan, Cyclophosphamide and Fludarabine
Brief Title: HSCT for Patients With Fanconi Anemia Using Risk-Adjusted Chemotherapy
Acronym: RAFA
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: Memorial Sloan Kettering Cancer Center (Other); Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-7501
Record Dates: First submitted 2014-04-28; First posted 2014-05-21 (Estimated); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Fanconi Anemia; Severe Marrow Failure; Myelodysplastic Syndrome (MDS); Acute Myelogenous Leukemia (AML)
Keywords: marrow aplasia; cytopenia; myelodysplasia; AML; bone marrow transplant; cytoreductive regimen; T-cell reduction
MeSH Terms: conditions — Fanconi Anemia; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute; Cytopenia; Anemia, Refractory, with Excess of Blasts | interventions — Busulfan; Cyclophosphamide; fludarabine; fludarabine phosphate; thymoglobulin; Granulocyte Colony-Stimulating Factor; Filgrastim; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Arm A: Good Risk Patients (Experimental): Patients 18 years old or younger with marrow aplasia or single lineage cytopenias will be receive intravenous busulfan (4 doses x 2 days), cyclophosphamide (4 doses x 4 days) and fludarabine (4 doses x 4 days), as used in our most current study that led to > 90% survival rates . Busulfan pharmacokinetics will not be used. All patients will receive rabbit ATG (4 doses x 4 days) prior to and granulocyte-colony stimulating factor (G-CSF) after transplant to promote engraftment. Cyclosporine will not be used for GVHD prophylaxis. The source of the stem cells for all patients will be peripheral blood stem cells mobilized by treatment of the donor with G-CSF. T-cell depletion will be performed by positive CD34 selection with the use of the Miltenyi system (CliniMACS device). Enrollment on this arm will include up to 50 patients.
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: rabbit ATG; Drug: G-CSF; Biological: Peripheral blood stem cell
- Arm B: Intermediate Risk Patients (Experimental): Patients 18 years old or younger with MDS or AML will receive intravenous busulfan (4 doses x 2 days), cyclophosphamide (4 doses x 4 days) and fludarabine (4 doses x 4 days). Busulfan pharmacokinetics will be used in this arm, as the dose of busulfan is higher. All patients will receive rabbit ATG (thymoglobulin) (4 doses x 4 days) prior to and G-CSF post transplant to promote engraftment. Cyclosporine will not be used for prophylaxis against GVHD. The source of the stem cells for all patients will be peripheral blood stem cells induced and mobilized by treatment of the donor. T-cell will be performed by positive CD34 selection with the use of the Miltenyi system (CliniMACS device).
  The maximum number of patients enrolled in this arm will be 10.
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: rabbit ATG; Drug: G-CSF; Biological: Peripheral blood stem cell
- Arm C: High Risk Patients (Experimental): Patients 19 years old or older with marrow aplasia or MDS or AML will receive intravenous busulfan (4 doses x 2 days), cyclophosphamide (4 doses x 4 days) and fludarabine (4 doses x 4 days). In this study, we will test whether outcomes can be improved, yet engraftment maintained, with a slightly reduced dose of busulfan. Patients will receive rabbit ATG (4 doses x 4 days) prior to and G-CSF post transplant to promote engraftment. Cyclosporine will not be used for GVHD prophylaxis. The source of the stem cells will be peripheral blood stem cells collected from donors treated with G-CSF. T-cell depletion will be performed by positive CD34 selection with the use of the Miltenyi system (CliniMACS device). The maximum number of patients enrolled will be 10.
  Interventions: Drug: Busulfan; Drug: Cyclophosphamide; Drug: Fludarabine; Drug: rabbit ATG; Drug: G-CSF; Biological: Peripheral blood stem cell

INTERVENTIONS:
Drug: Busulfan — A standard dose of busulfan, associated with excellent outcomes in our previous trial will be used for young patients with marrow aplasia (arm A).
  A higher dose of busulfan will be used in younger patients with MDS and AML (arm B) to maximize disease control.
  A lower dose of busulfan will be used in older patients (arm C) to minimize toxicity.
  Other Names: Myleran; Busulfex IV
Drug: Cyclophosphamide — Arms A, B and C - Cytoxan will be given as a 1-2 hour infusion for 4 days. The dose will be adjusted according to patients ideal body weight for obese patients.
  Other Names: Cytoxan
Drug: Fludarabine — Arms A, B and C - Fludarabine will be given IV over 30 minutes daily for 4 days. The dose will be adjusted according to renal function according to Institutional guidelines.
  Other Names: Fludara
Drug: rabbit ATG — Arms A, B and C - 4 doses will be given prior to transplant to promote engraftment.
  Other Names: thymoglobulin
Drug: G-CSF — All patients will also receive G-CSF post-transplant to foster engraftment.
  Other Names: Granulocyte colony-stimulating factor; filgrastim; neupogen
Biological: Peripheral blood stem cell — The source of stem cells for all patients will be peripheral blood stem cells (PBSC) induced and mobilized by treatment of the donor with G-CSF for 4-6 days. T-cell depletion will be uniformly performed by positive CD34 selection with the use of the Miltenyi system (CliniMACS device).

SUMMARY:
The purpose of this study is to determine whether the use of lower doses of busulfan and the elimination of cyclosporine will further reduce transplant-related side effects for patients with Fanconi Anemia (FA). Patients will undergo a transplant utilizing mis-matched related or matched unrelated donors following a preparative regimen of busulfan, fludarabine, anti-thymocyte globulin and cyclophosphamide.

DETAILED DESCRIPTION:
The trial proposed is a three arm phase II treatment protocol designed to investigate the safety and efficacy of risk-adjusted chemotherapy-based cytoreductive regimen plus a CD34+ selected T-cell depleted peripheral blood stem cell (PBSC) stem cell transplant for the treatment of patients with Fanconi anemia and severe hematologic disease. Candidates for this trial will include patients with Fanconi anemia presenting with severe marrow failure (transfusion dependent) or myelodysplastic syndrome, or acute myelogenous leukemia for whom an allogeneic stem cell transplant is indicated.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have a diagnosis of Fanconi anemia
* Patients must have one of the following hematologic diagnoses:

  1. Severe Aplastic Anemia (SAA), with bone marrow cellularity of <25% OR Severe Isolated Single Lineage Cytopenia and at least one of the following features:

     1. Platelet count <20 x 109/L or platelet transfusion dependence*
     2. ANC <1000 x 109/L
     3. Hgb <8 gm/dl or red cell transfusion dependence*
  2. Myelodysplastic Syndrome (MDS) (based on WHO or IPSS Classification
  3. Acute Myelogenous Leukemia (untreated, in remission or with refractory or relapsed disease)
* Donors will be either human leukocyte antigen (HLA) compatible unrelated or HLA-genotypically matched related donors (no fully matched sibling donor).
* Patients and donors may be of either gender or any ethnic background.
* Patients must have a Karnofsky adult, or Lansky pediatric performance scale status > 70%.
* Patients must have adequate physical function measured by:

  1. Cardiac: asymptomatic or if symptomatic then 1) left ventricular ejection fraction (LVEF) at rest must be > 50% and must improve with exercise or 2) Shortening Fraction > 29%
  2. Hepatic: < 5 x upper limit of normal (ULN) alanine transaminase (ALT) and < 2.0 mg/dl total serum bilirubin.
  3. Renal: serum creatinine <1.5 mg/dl or if serum creatinine is outside the normal range, then CrCl > 50 ml/min/1.73 m2
  4. Pulmonary: asymptomatic or if symptomatic, DLCO > 50% of predicted
* Each patient must be willing to participate as a research subject and must sign an informed consent form.
* Female patients and donors must not be pregnant or breastfeeding at the time of signing consent. Women must be willing to undergo a pregnancy test prior to transplant and avoid becoming pregnant while on study.

Exclusion Criteria:

* Active CNS leukemia
* Female patients who are pregnant (positive serum or urine HCG) or breast-feeding.
* Active uncontrolled viral, bacterial or fungal infection
* Patient seropositive for HIV-I/II; HTLV -I/II

Min Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2014-04; Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Graft Failure or Rejection | 5 years
  Primary non-engraftment is diagnosed when the patient fails to achieve an ANC >=500/mm3 at any time in the first 28 days post-transplant. If (1) after achievement of an absolute neutrophil count (ANC) >=500/mm3, the ANC declines to <500/mm3 for more than 3 consecutive days in the absence of relapse, or, (2) there is absence of donor cells in the marrow and/or blood as demonstrated by chimerism assay in the absence of relapse, a diagnosis of secondary graft failure is made. The patient is not evaluable for graft failure or rejection if recurrence of host MDS is detected concurrently.

SECONDARY OUTCOMES:
Post-transplant severe morbidity and mortality | 2 years post-transplant
  The occurrence of severe post-transplant regimen-related severe morbidity (grade IV toxicity) and/or mortality will be the second endpoint of this study. In the context of the agents or agent-combination used for cytoreduction used, particular attention will be given to toxicity involving (1) the liver, (2) the lungs, (3) the oral mucosa and gastrointestinal tract, and (4) the central nervous system.

OTHER OUTCOMES:
Graft Versus Host Disease | One year
  Patients will be observed for acute and/or chronic graft versus host disease (GvHD). Standard clinical criteria for the grading of acute and chronic GvHD will be done according to IBMTR guidelines.
Leukemic Relapse | 5 years
  For patients with MDS or AML, relapse will be analyzed as to type and genetic origin of the MDS/leukemic cells.
Secondary malignancies | 5 years
  Patients will be followed for 5 years through annual contact with their treatment center in order to track the risk of developing a secondary malignancy.

CONTACTS AND LOCATIONS:
Overall Officials: Parinda Mehta, MD, Principal Investigator — CCHMC
Locations (3):
- United States (3):
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Fred Hutchinson Cancer Research Center, Seattle, Washington